CLINICAL TRIAL: NCT05106933
Title: The Effect of Carbohydrate Loading 2 Hours Before Upper Endoscopy on Gastric Residual Volume and Patient's Well-being Score : A Single-Blind, Randomized Controlled Trial Study
Brief Title: The Effect of Carbohydrate Loading 2 Hours Before Gastroscopy on Gastric Residual Volume and Patient's Well-being Score
Acronym: Carborie
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, MOHD FIRDAUS BIN ZULKIFLI, Dr. Mohd Firdaus bin Zulkifli, Hospital Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HUSM Malaysia
Record Dates: First submitted 2021-10-09; First posted 2021-11-04 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Gastric Residual Volume; Upper Endoscopy
Keywords: GRV

STUDY DESIGN:
Intervention Model Description: Carbohydrate loading vs Clear water
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plain water (Placebo Comparator): Group A patient will be given 400cc of plain water, 2 hours prior to gastroscopy
  Interventions: Other: Plain water
- Carborie (Experimental): Group B patient will be given 400cc of carborie (carbohydrate drink), 2 hours prior to gastroscopy
  Interventions: Other: Carborie

INTERVENTIONS:
Other: Plain water — Measure gastric residual volume during upper endoscopic, after given plain water and carborie 2 hours prior upper endoscopy
  Arms: Plain water
Other: Carborie — carbohydrate drink
  Arms: Carborie

SUMMARY:
This is a single-blind randomized controlled trial with a stratified (diabetes mellitus, non-diabetes mellitus), balanced randomization (1:1), placebo-controlled study regarding the effect of carbohydrate loading 2 hours prior to the outpatient upper endoscopic procedure. All patients who were assigned for outpatient oesophagogastroduodenoscopy (OGDS) were invited to join in this study voluntarily from January 2021 until August 2021. This study was conducted in the Endoscopy Unit, Hospital Universiti Sains Malaysia, Kubang Kerian, Malaysia. The endoscopists that performed this procedure were blinded and there was trained staff who was not involved in the study to assess the well-being score. The study protocol had been approved by the Human Research Ethics Committee of Universiti Sains Malaysia (JEPeM) with the assigned protocol code USM/JEPeM/20080414.

DETAILED DESCRIPTION:
Patient planned for OGDS in HUSM will be randomized into 2 groups. Plain water is given to group A of subject and carbohydrate loading is given to group B subject 2 hours before OGDS. Gastric residual volume is visualized directly and measured through aspiration via OGDS and subject's well-being is assessed for both group of the subject prior and after clear fluid have been given.

Methodology :

Research design :- This is a single-blind randomized controlled trial. This is a stratified (diabetes mellitus, non-diabetes mellitus) with balanced randomization (1:1), placebo-controlled study Study area :- This study will be conducted in the endoscopy room, Hospital Universiti Sains Malaysia (HUSM) in Kubang Kerian, Kelantan, Malaysia

All subjected planned for OGDS with the complaint of one or more of the following symptoms : Bothersome postprandial fullness, early satiety, epigastric pain or epigastric burning and fulfill the inclusion criteria are selected. Patients will be approached and be explained regarding the study in surgical outpatient clinic before OGDS. The patient will be approached again on the day of OGDS, if agree to participate, informed consent will be obtained. Informed consent will be obtained after explanation regarding the study and procedure again by researcher nurse.

The allocation sequence is according to computer-generated random number list, it was prepared by an investigator with no clinical involvement in the trial. The allocation sequence was concealed from researcher enrolling and assessing participants. The allocation sequence will be sealed in sequentially numbered and opaque envelopes. A manila card will be placed inside envelop to render it impermeable to intense light. To prevent subversion of the allocation sequence, the name and identification number of the participants will be written on a book together with the series number on the envelope. The details in the book will be kept confidentially.

After enrolled subject complete all the baseline assessment, the corresponding envelope will be enclosed by the trained staff (who not involved in the study) who prepare the drink. The staff need to ensure that the envelop is still sealed when receiving it. The staff will prepare the drink into an identical container according to the assignment.

The subjects are randomized into 2 groups: 1 group with 400mL plain water and another group given 1 packet carborie (400mL). Subjects need to finish the drink over 10 minutes. After that, subjects are not allowed to leave endoscope room until finish OGDS to prevent consumption of other drink or food.

2 hours after that, the subject undergoes OGDS. OGDS is performed following the standard protocol.

1. The patient lies in the left lateral position
2. Medication/lignocaine spray to numb the back of throats (spray) will be given to prevent gagging during the passage of the instrument
3. A plastic mouth guard (mouthpiece) is placed between the teeth to prevent damage to the teeth and endoscope
4. The endoscope (also called a gastroscope) will be inserted through the mouthpiece
5. A small container or yankauer suction is placed close to the mouth of a patient to collect saliva during and after the oesophagogastroduodenoscopy (OGDS)
6. The endoscope will be inserted along the middle line of the soft palate
7. Once endoscope advanced, the patient may be asked to swallow to facilitate advancement of scope
8. Throughout the procedure, no water flushing is allowed, only air inflation is allowed.

Visualized pooling of fluid in the stomach is aspirated until dry via direct visualization with the endoscope. The aspirated fluid will be collected in the suction reservoir and the fluid will be measured

Subject's well-being score is assessed via visual analogue scale (VAS) which consist of 5 parameters: hunger, thirst, anxiety, tiredness and general discomfort. This scale will be used repeatedly during this study to assess the patient's well-being. The trained staff nurse will ask the patient regarding the level of 5 parameters and subject need to mark [X] somewhere along the horizontal line given before drink and before OGDS procedure.

All subjects are advised to inform assessor if there is an adverse reaction. Medical personnel are available to manage any adverse events that might occur throughout the procedure.

The possible risk that may arise in the study includes injury to the gastrointestinal wall, aspiration and bleeding which is the similar risk for all patient undergoing for OGDS procedure. The small volume of the drink will not cause psychological distress to the subject, but its taste may not be palatable.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years old and above
* Agree to participate

Exclusion Criteria:

* History of upper gastrointestinal surgery
* Patient with active gastrointestinal bleeding
* Unstable clinical condition
* Mentally disable or who cannot give an informed consent
* Patient on the nasogastric feeding tube
* Pregnant patient
* American Society of Anesthesiologists classification of physical status grade 3 or above
* Insulin dependent Diabetes Mellitus more than 10 years
* Patient who is carbohydrate intolerance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-10-20 (Actual)

PRIMARY OUTCOMES:
To compare the gastric residual volume 2 hours after carbohydrate loading (intervention group) and plain water group (control group) | 2 hour before OGDS
  Patients will be randomised into control group and intervention group. Those in intervention group will have to drink clear water containing carbohydrate (carborie) 2 hours prior to gastroscopy. Endoscopist will measure patient's gastric residual volume. Residual gastric fluid will be aspirated into the container, final volume will be measured.

SECONDARY OUTCOMES:
To compare the patient's well-being after ingestion of carbohydrate loading (intervention group) and plain water (control group) | 2 hours
  To assess patient well-being score before and after giving carborie load. Visual analogue scale (VAS) used for assessment of patient well-being. Just before and after the ingestion of the clear fluid patients are told to indicate the level of discomfort on a visual analogue scale which ranged from 0mm to 100mm. Zero signifying not at all while 100 signify the most imaginable/maximum discomfort.

OTHER OUTCOMES:
To assess the effect of carbohydrate loading in patient planned for OGDS in HUSM | 2 hours prior OGDS
  To assess gastric residual volume 2 hour prior OGDS

CONTACTS AND LOCATIONS:
Overall Officials: Nizam Hashim, Master, Study Director — HUSM, Kubang Kerian, Malaysia
Locations (1):
- Department of General Surgery, Kota Bharu, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Qureshi WA, Zuckerman MJ, Adler DG, Davila RE, Egan JV, Gan SI, Lichtenstein DR, Rajan E, Shen B, Fanelli RD, Van Guilder T, Baron TH; Standards of Practice Committee, American Society for Gastrointestinal Endoscopy. ASGE guideline: modifications in endoscopic practice for the elderly. Gastrointest Endosc. 2006 Apr;63(4):566-9. doi: 10.1016/j.gie.2006.02.001. No abstract available. PMID 16564853
- [Result] De Silva AP, Amarasiri L, Liyanage MN, Kottachchi D, Dassanayake AS, de Silva HJ. One-hour fast for water and six-hour fast for solids prior to endoscopy provides good endoscopic vision and results in minimum patient discomfort. J Gastroenterol Hepatol. 2009 Jun;24(6):1095-7. doi: 10.1111/j.1440-1746.2009.05782.x. Epub 2009 Feb 12. PMID 19220672
- [Result] Sabry R, Hasanin A, Refaat S, Abdel Raouf S, Abdallah AS, Helmy N. Evaluation of gastric residual volume in fasting diabetic patients using gastric ultrasound. Acta Anaesthesiol Scand. 2019 May;63(5):615-619. doi: 10.1111/aas.13315. Epub 2019 Jan 4. PMID 30609007
- [Result] Spada C, McNamara D, Despott EJ, Adler S, Cash BD, Fernandez-Urien I, Ivekovic H, Keuchel M, McAlindon M, Saurin JC, Panter S, Bellisario C, Minozzi S, Senore C, Bennett C, Bretthauer M, Dinis-Ribeiro M, Domagk D, Hassan C, Kaminski MF, Rees CJ, Valori R, Bisschops R, Rutter MD. Performance measures for small-bowel endoscopy: A European Society of Gastrointestinal Endoscopy (ESGE) Quality Improvement Initiative. United European Gastroenterol J. 2019 Jun;7(5):614-641. doi: 10.1177/2050640619850365. Epub 2019 May 15. PMID 31210941
- [Result] American Society of Anesthesiologists Committee. Practice guidelines for preoperative fasting and the use of pharmacologic agents to reduce the risk of pulmonary aspiration: application to healthy patients undergoing elective procedures: an updated report by the American Society of Anesthesiologists Committee on Standards and Practice Parameters. Anesthesiology. 2011 Mar;114(3):495-511. doi: 10.1097/ALN.0b013e3181fcbfd9. No abstract available. PMID 21307770
- [Derived] Zulkifli MF, Md Hashim MN, Zahari Z, Wong MP, Syed Abd Aziz SH, Yahya MM, Wan Zain WZ, Zakaria AD, Ramely R, Jien Yen S, Othman MF. The effect of pre-endoscopy maltodextrin beverage on gastric residual volume and patient's well-being: a randomised controlled trial. Sci Rep. 2023 Nov 16;13(1):20078. doi: 10.1038/s41598-023-47357-5. PMID 37973795